CLINICAL TRIAL: NCT05146362
Title: One-Year Impact Evaluation of Vermont Retaining Employment and Talent After Injury/Illness Network (RETAIN)
Brief Title: Vermont RETAIN Impact Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Social Security Administration (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RTN-VT; OD-36366-21-75-4-50 (Other Grant/Funding Number: Social Security Administration)
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Disability
Keywords: disability; unemployment; employment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RETAIN Programming (Experimental): The experimental group receives the full set of RETAIN intervention activities.
  Interventions: Other: Vermont RETAIN
- Control (No Intervention): This arm receives information about American Job Center services and assistance with opening a JobLink account if an individual doesn't have one. Medical providers at all practices will receive training on how to identify early and then manage the risk of work disability to help prevent long-term unemployment

INTERVENTIONS:
Other: Vermont RETAIN — RETAIN projects include a combination of medical provider services, stay-at-work/return-to-work (SAW/RTW) coordination services, and other SAW/RTW services. The evaluation compares the treatment group that is eligible to receive the full set of RETAIN intervention activities and a control group that is not.
  Arms: RETAIN Programming

SUMMARY:
The Retaining Employment and Talent after Injury/Illness Network (RETAIN) demonstration is a collaborative effort between the U.S. Department of Labor (DOL) and the Social Security Administration (SSA) to improve employment outcomes for individuals who experience injuries or illnesses that put them at risk of exiting the labor force and relying on disability programs and other public supports in the long term. RETAIN projects include a combination of medical provider services, stay-at-work/return-to-work (SAW/RTW) coordination services, and other SAW/RTW services. This evaluation will focus on the Vermont Department of Labor's implementation of "Vermont RETAIN" statewide. The evaluation will document how the project is implemented, describe enrollees, estimate the project's impacts on enrollees' outcomes, and assess whether the benefits outweigh the costs.

DETAILED DESCRIPTION:
The Vermont Department of Labor is partnering with health care, employment, and other entities to implement "Vermont RETAIN." SSA contracted with Mathematica to conduct an independent evaluation of the program. Under the RETAIN model medical providers receive training and incentives to use occupational health best practices. The state agency also coordinates SAW/RTW services for the enrollee, fosters communication among Vermont RETAIN stakeholders about the treatment enrollee returning to work, and monitors the enrollee's medical and employment progress. Providers at participating practices are trained in the Vermont Best Practice Resources and Training, which explains how to identify early and then manage the risk of work disability to help prevent long-term unemployment. Participants undergo a systematic assessment of barriers to work, work goals, and function in order to create a personalized RTW plan; RTW coordinators use a strength-based coaching model and provide care coordination through a customized mobile health app.

Vermont plans to work with 68 primary care practices across the state and enrolls clusters of medical practices to participate in the study. The evaluation team randomly assigns each cluster to either a treatment or control group. Mathematica conducts random assignment of clusters on a rolling basis as Vermont enrolls clusters. Vermont invites eligible individuals who see a medical provider in either the treatment or control group to enroll in the study. Individuals who see a provider that has been randomly assigned to the treatment group and who enroll in the study are considered "treatment group enrollees" and are eligible for Vermont RETAIN services. Individuals who see a provider in the control group and enroll in the study are considered "control group enrollees" and are not eligible for Vermont RETAIN services.

The evaluation team then compares the outcomes of the treatment and control groups and gathers evidence on how RETAIN shaped the outcomes of enrollees who were eligible for its services, regardless of whether they participated in those services. Data sources include enrollment data, surveys, administrative records, program data, and qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Live or work in Vermont (or if out of work, lives in a border state and plan to work in Vermont)
* Currently employed or actively looking for a job
* Have an injury or illness that is limiting or could limit ability to stay at or return to work
* The injury or illness occurred, flared, or worsened within the past 6 months

Exclusion Criteria:

* Has received care of coordination services from RETAIN before
* Has an active SUD that is currently untreated
* Has been out of work for more than 12 weeks due to injury, illness, or flare
* Currently applying for or receiving disability benefits from Social Security Administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2040 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Share of enrollees employed in the fourth quarter after enrollment | Measured in the fourth quarter after enrollment
  Share of enrollees employed in the fourth quarter after enrollment obtained from state unemployment insurance wage records. These files include individual-level wage records for six quarters surrounding enrollment in the study, including the quarter prior to enrollment, the quarter of enrollment, and four post-enrollment quarters.
Enrollee earnings in the fourth quarter after enrollment | Measured in the fourth quarter after enrollment
  Sum of enrollee earnings in the fourth quarter after enrollment obtained from state unemployment insurance wage records. These files include individual-level wage records for six quarters surrounding enrollment in the study, including the quarter prior to enrollment, the quarter of enrollment, and four post-enrollment quarters.
Share of enrollees that applied for SSDI or SSI during the 12 months after enrollment | Measured in the 12 months after enrollment
  Share of enrollees that applied for SSDI or SSI during any of the 12 months after enrollment obtained from SSA program data. These files include detailed information about Social Security Disability Insurance (SSDI) and Supplemental Security Income (SSI) applications SSDI and SSI awards, SSDI and SSI benefit amounts and enrollee characteristics (for enrollees who have ever applied for SSA program benefits)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Berk, PhD, Principal Investigator — Mathematica Policy Research, Inc.
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No